CLINICAL TRIAL: NCT04009655
Title: The Effects of Music Therapy on Near-infrared Spectroscopy and Electroencephalogram in Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MTOBF
Record Dates: First submitted 2019-05-31; First posted 2019-07-05 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Preterm Infant; Music; Near-infrared Spectroscopy; Electroencephalogram
MeSH Terms: conditions — Premature Birth | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- music therapy (Experimental): The infant will receive music therapy over 3 consecutive days and will obtain standard care as usual
  Interventions: Other: music
- control (No Intervention): The infant does not receive any sound emission because the headphone will be turned off and will obtain standard care as experimental

INTERVENTIONS:
Other: music — music selected by musician
  Arms: music therapy

SUMMARY:
Music has been consistently shown magic power in brain plasticity. Several study proved music can influence electronic activity of preterm infants' brain, while none study covered region oxygen metabolic. The investigators aim to discover the effects of music therapy on near-infrared spectroscopy and electroencephalogram in premature infants.

DETAILED DESCRIPTION:
Previous studies of music therapy have made some achievements for adult Parkinson's disease, schizophrenia, depression, anxiety, post-traumatic stress and pediatric autism spectrum disorders. For newborns, studies mainly focused on the effects of basic vital signs, feeding and pain score decreasing. So far, no studies evaluating the effect of music therapy on brain oxygen metabolic and electronic activity.

ELIGIBILITY:
Inclusion Criteria:

* Postmenstrual age of 32-36+6 weeks.
* Appropriate weight for gestational age.
* To have signed an informed consent to participate in the study.
* Have reached clinical stability.

Exclusion Criteria:

* Have nervous system diseases or obvious nervous system symptoms.
* Severe congenital diseases.
* The maintenance of sedative or analgesic drugs.
* Support with mechanical ventilation.

Ages: 224 Days to 258 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
change of brain oxygen saturation | from the start of the intervention to the end of the 3rd day
  near-infrared spectroscopy to monitor brain oxygen saturation

SECONDARY OUTCOMES:
Burdjalov Scores of amplitude integrated electroencephalogram | from the start of the intervention to the end of the 3rd day
  electroencephalogram to monitor brain electronic activity, using Burdjalov developed cerebral function monitoring scoring system which including: (1)record continuity: assessed through observing the overall density of the sample tracing, scores ranged from 0 to 2；(2) presence of cyclic changes：refers to the emergence and progression of periods during monitoring，scores ranged from 0 to 5；（3）degree of voltage amplitude depression：estimated as the average lower microvolt level during the recording epoch ，scores ranged from 0 to 2；（4）bandwidth：reflects a combination of the voltage span (peak-to-trough) of the tracing and the magnitude of the electroencephalogram depression，scores ranged from 0 to 4. The minimum possible total score was 0, and the maximum was 13. Scores progressively increased with central nerve system maturation.
change of heart rates | from the start of the intervention to the end of the 3rd day
  monitors recording heart rates
change of respiratory rates | from the start of the intervention to the end of the 3rd day
  monitors recording respiratory rates
change of pluse oxygen saturation | from the start of the intervention to the end of the 3rd day
  monitors recording transcutaneous oxygen saturation

CONTACTS AND LOCATIONS:
Overall Officials: lai s wang, Ph.D, Study Director — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China